CLINICAL TRIAL: NCT02290379
Title: A Single-Center, Randomized, Double-blind, Placebo-controlled, Phase 1, Single Ascending Dose Safety, Tolerability, and Pharmacokinetic Study of TNX-201 Capsules in Healthy Volunteers.
Brief Title: Phase 1 Single Ascending Dose Safety Study of TNX-201 Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TNX-IS-T101
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2014-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- TNX-201 35 mg (Experimental): Drug: TNX-201 35 mg
  Interventions: Drug: TNX-201 35 mg
- TNX-201 70 mg (Experimental): Drug: TNX-201 70 mg
  Interventions: Drug: TNX-201 70 mg
- TNX-201 140 mg (Experimental): Drug: TNX-201 140 mg
  Interventions: Drug: TNX-201 140 mg
- Racemic isometheptene 70 mg (Active Comparator): Comparator: Racemic Isometheptene 70 mg
  Interventions: Drug: Racemic isometheptene 70 mg
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNX-201 35 mg — Drug: TNX-201 35 mg
  Arms: TNX-201 35 mg
Drug: TNX-201 70 mg — Drug: TNX-201 70 mg
  Arms: TNX-201 70 mg
Drug: TNX-201 140 mg — Drug: TNX-201 140 mg
  Arms: TNX-201 140 mg
Drug: Racemic isometheptene 70 mg — Active Comparator: Racemic isometheptene 70 mg
  Arms: Racemic isometheptene 70 mg
Drug: Placebo — Drug: Placebo
  Arms: Placebo

SUMMARY:
Single-center, randomized, double-blind, placebo-controlled, single ascending dose, safety and tolerability study of TNX-201 capsules in healthy volunteers.

DETAILED DESCRIPTION:
Single-center, randomized, double-blind, placebo-controlled, single ascending dose, safety and tolerability study of TNX-201 capsules in healthy volunteers. Three successive cohorts are planned with doses of TNX-201 capsules, 35 mg, 70 mg, and 140 mg, respectively. Each cohort will consist of 15 subjects, and subjects will be randomly assigned to TNX-201, racemic isometheptene, or placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 and ≤ 55 years of age on the day of randomization. NOTE: At least 6 female subjects need to be randomized in each cohort.
2. Body mass index (BMI) ≥18.5 and ≤33.0
3. Non-tobacco users (no use of tobacco- or nicotine- containing products within 3 months prior to study drug administration)

Exclusion Criteria:

1. Any clinically significant abnormality or clinically significant abnormal laboratory test results found at Screening or Day -1, or a positive test for HBsAg, HCAb, or HIV found at Screening
2. Positive urine drug screen (including alcohol, tetrahydrocannabinol (THC), cocaine, amphetamines, and opiates) or urine cotinine test at Screening or on Day -1
3. Known or suspected hypersensitivity to isometheptene mucate or any excipients used in the formulations.
4. Positive serum pregnancy test at Screening or Day -1
5. Any reason, in the opinion of the Principal Investigator (PI) or the sponsor's Medical Monitor, to prevent the subject from participating in the study
6. Clinically significant ECG abnormalities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Plasma levels of isometheptene or metabolites. | 60 minutes pre-dose and multiple timepoints up to 48 hours post-dose
Number of Adverse events | 60 minutes pre-dose and multiple timepoints up to 48 hours post-dose